CLINICAL TRIAL: NCT03479645
Title: Can a Multimodal Approach Using SMS Reminders and an Opt-out Mailed FIT Kits Improve Participation in Colorectal Cancer Screening? A Single Center Randomized Controlled Trial
Brief Title: Serial SMS Reminders and an Opt-out Mailed FIT Kits to Improve Colorectal Screening Participation: A Single Center RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 828624
Record Dates: First submitted 2018-02-23; First posted 2018-03-27 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Bowel Cancer; Colon Cancer
Keywords: Colon cancer; Bowel cancer; Cancer screening; text message; Fecal immunochemistry test (FIT); opt-out; behavioral intervention
MeSH Terms: conditions — Intestinal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control arm - usual practice. Simple SMS reminder that informs patients they are overdue for CRC screening and requests they contact the clinic.
- Intervention (Experimental): Serial text messages and mailed FIT kit
  Interventions: Behavioral: Serial text messages and mailed FIT kit

INTERVENTIONS:
Behavioral: Serial text messages and mailed FIT kit — 1. Pre-alert SMS offering Opt-out of mailed FIT kit
  2. Mailed home FIT kit
  3. SMS A - Reciprocity message
  4. SMS B - Offer for second FIT kit if lost/did not receive
     * Plus SMS A + C if second mailed FIT is requested.
  5. SMS C - Salience message
  Arms: Intervention

SUMMARY:
This pilot study is a 2-armed randomized controlled trial assessing the impact of a multimodal approach on colorectal cancer screening participation rates in a Federally Qualified Health Center. The trial will test serial text message reminders and opt-out mailed fecal immunochemistry test (FIT) home kits against a simple reminder text message control. Patients aged 50-74 years, who are registered at a Family Practice and Counselling Network (FPCN) clinic and are overdue for colorectal cancer screening will be recruited. The primary outcome is the rate of FIT kits being returned at 12 weeks.

DETAILED DESCRIPTION:
It is estimated that colorectal cancer (CRC) screening can reduce the risk of dying from bowel cancer by approximately 15%. Yet despite this, the national participation rate is only approximately 62.9%, highlighting that the national target of 70.5% set out in the Healthy People 2020 Objectives remains well out of reach. The US Preventative Task Force (USPSTF) recommends colorectal screening for adults aged 50-75 years through either annual fecal occult blood testing (FOBT), flexible sigmoidoscopy every 5 years or colonoscopy every 10 years. However, many service providers rely on the opportunistic offer of screening at existing health touch-points. This requires the patient to see their healthcare provider, usually for a different clinical reason, the provider to recognize that the patient is overdue for CRC screening and the provider to recommend and book the patient for CRC screening. This process identifies a number of barriers encountered at the system, provider and patient level, to completing a screening test regularly. Furthermore, much evidence indicates that public participation in colorectal screening is heavily influences by socioeconomic factors. Lower participation rates are seen in individuals without health insurance, without a medical home, who are more deprived and from ethnic minority groups. These individuals are more likely to present with later stage disease and experience poorer outcomes. Fecal immunochemistry testing (FIT) is a stool sample based test kit that uses antibodies to detect the human haemoglobin protein in the stool sample and can be completed in the privacy of the home. Research has showed that mailed home test kits such as FOBT or FIT kits can improve CRC participation by reducing the effort required to see a provider in order to arrange CRC screening. Evidence has also shown that text message reminders can improve participation in cancer screening. Furthermore, the message content of text messages can differentially change behavior, for example reducing the 'did not attend rate' in hospital outpatient appointments but also in the context of participation in cervical cancer screening. Therefore this trial will test a multimodal outreach approach, which uses serial SMS reminders with different word contents and mailed FIT kits on the participation rates of CRC screening.

ELIGIBILITY:
Inclusion Criteria:

1. aged 50-74
2. at least 1 clinic visit to the FPCN within the previous 12 months
3. due or overdue for colorectal screening
4. Asymptomatic for bowel cancer
5. mobile phone number available

Exclusion Criteria:

1. Has had prior colonoscopy within 10 years, sigmoidoscopy within 5 years, and FOBT/FIT within twelve months of the chart review (We will exclude patients who self-report undergoing any of the above procedures)
2. Has a history of CRC
3. Has a history of other GI cancer
4. Has history of confirmed Inflammatory Bowel Disease (IBD) (e.g. Crohns disease, ulcerative colitis) Irritable bowel syndrome does not exclude patients.
5. Has history of colitis other than Crohns disease or ulcerative colitis
6. Has had a colectomy
7. Has been diagnosed with Lynch Syndrome (i.e. HNPCC)
8. Has been diagnosed with Familial Adenomatous Polyposis (FAP)
9. Has metastatic (Stage IV) blood or solid tumor cancer
10. Has end stage renal disease
11. Has dementia
12. Has liver cirrhosis
13. Has any other condition that, in the opinion of the investigator, excludes the patient from participating in this study.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
Colorectal screening rate | 12 weeks
  The rate patients with who completed colorectal screening within the trial period

SECONDARY OUTCOMES:
Per Protocol analysis: Colorectal screening rate | 12 weeks
  The rate of FIT kit return by trial arm in individuals who received at least the first text message, who did not self-report being up to date with colorectal cancer screening.
FIT kit return rate | 12 weeks
  The rate of FIT kit return by trial arm
Per protocol analysis: FIT kit return rate | 12 weeks
  The rate of FIT kit return by trial arm, in participants who received at least the first text message, who did not self-report being up to date with colorectal cancer screening.
colonoscopy completion rate | 12 weeks
  The rate of colonoscopy within the trial period by trial arm
Per protocol analysis: colonoscopy completion rate | 12 weeks
  The rate of colonoscopy within the trial period by trial arm, in participants who received at least the first text message, who did not self-report being up to date with colorectal cancer screening.
Colorectal screening return rate by gender | 12 weeks
  Uptake of screening and FIT return by gender
FIT return rate by gender | 12 weeks
  Uptake of screening and FIT return by gender
Colorectal screening rate by insurance status | 12 weeks
  Uptake of screening by insurance status
FIT kit return rate by insurance status | 12 weeks
  FIT return by insurance status

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Family Practice and Councelling Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardcastle JD, Chamberlain JO, Robinson MH, Moss SM, Amar SS, Balfour TW, James PD, Mangham CM. Randomised controlled trial of faecal-occult-blood screening for colorectal cancer. Lancet. 1996 Nov 30;348(9040):1472-7. doi: 10.1016/S0140-6736(96)03386-7. PMID 8942775
- [Background] Halpern MT, Ward EM, Pavluck AL, Schrag NM, Bian J, Chen AY. Association of insurance status and ethnicity with cancer stage at diagnosis for 12 cancer sites: a retrospective analysis. Lancet Oncol. 2008 Mar;9(3):222-31. doi: 10.1016/S1470-2045(08)70032-9. Epub 2008 Feb 20. PMID 18282806
- [Background] Clegg LX, Li FP, Hankey BF, Chu K, Edwards BK. Cancer survival among US whites and minorities: a SEER (Surveillance, Epidemiology, and End Results) Program population-based study. Arch Intern Med. 2002 Sep 23;162(17):1985-93. doi: 10.1001/archinte.162.17.1985. PMID 12230422
- [Background] Institute NC. Caner trends progress reprot; Colorectal Screening. https://progressreport.cancer.gov/detection/colorectal_cancer
- [Background] von Wagner C, Baio G, Raine R, Snowball J, Morris S, Atkin W, Obichere A, Handley G, Logan RF, Rainbow S, Smith S, Halloran S, Wardle J. Inequalities in participation in an organized national colorectal cancer screening programme: results from the first 2.6 million invitations in England. Int J Epidemiol. 2011 Jun;40(3):712-8. doi: 10.1093/ije/dyr008. Epub 2011 Feb 17. PMID 21330344
- [Background] Power E, Miles A, von Wagner C, Robb K, Wardle J. Uptake of colorectal cancer screening: system, provider and individual factors and strategies to improve participation. Future Oncol. 2009 Nov;5(9):1371-88. doi: 10.2217/fon.09.134. PMID 19903066
- [Derived] Huf SW, Asch DA, Volpp KG, Reitz C, Mehta SJ. Text Messaging and Opt-out Mailed Outreach in Colorectal Cancer Screening: a Randomized Clinical Trial. J Gen Intern Med. 2021 Jul;36(7):1958-1964. doi: 10.1007/s11606-020-06415-8. Epub 2021 Jan 28. PMID 33511567